CLINICAL TRIAL: NCT02621801
Title: Evaluation of a Mind-body Education Program to Enhance Resiliency and Reduce Burnout in Residents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: NYU Langone Health (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, John W. Denninger, MD, PhD, Principle Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015P000916
Record Dates: First submitted 2015-11-23; First posted 2015-12-04 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Resident Burnout

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Stress Management and Resiliency Training for Residents (SMART-R)
  Interventions: Behavioral: Stress Management and Resiliency Training for Residents (SMART-R)
- Waitlist Control (Active Comparator): The control group will receive the same intervention (SMART-R) after the experimental group.
  Interventions: Behavioral: Stress Management and Resiliency Training for Residents (SMART-R)

INTERVENTIONS:
Behavioral: Stress Management and Resiliency Training for Residents (SMART-R) — The Stress Management and Resiliency Training Program for residents (SMART-R) is a six-hour intervention delivered over 2 or 3 sessions that teaches residents mind-body skills to reduce stress and enhance coping strategies.

SUMMARY:
This prospective, waitlist-control study is evaluating the benefits of a stress management and resiliency training program for residents (SMART-R).

The primary aim of this study is to determine whether the SMART-R is effective at increasing coping skills and reducing stress among residents, reflected by changes in constructs such as emotional growth, perceived stress, optimism, and coping styles. Objective parameters (heart rate, galvanized skin response, sleep duration and quality, exercise and actigraphy) measured with the Basis health tracking device will help correlate objective signs to subjective report of stress.

DETAILED DESCRIPTION:
The investigators adapted the Benson-Henry Institute Stress Management and Resiliency Training Program -- Relaxation Response Resiliency Program (SMART-3RP) to create the SMART-R resident wellness curriculum. The actual SMART-3RP is both a clinical program and research intervention. The three prongs of the SMART-R include 1) elicitation of the relaxation response through mind-body techniques 2) reducing overall stress reactivity and 3) increasing connectedness to self and others.

In a waitlist-control design, the SMART-R was implemented into multiple residents programs at Mass General Hospital, NYU Langone Medical Center, and Weill Cornell Medical College. The primary aim is to evaluate the effectiveness of the SMART-R in increasing coping skills and reducing stress among residents in the participating programs. Participants enrolled will be invited to complete 1) a brief questionnaire before, during (q3months) and after participation in the program (5 questionnaires total). The investigators will also collect continuous physiologic data using the Basis Peak Health Tracking device to correlate the physiologic data with self-report measures of stress.

Additionally, objective indicators of daily workload (page frequency, and quantity of notes authored by a resident during a given period) will help control for residents' schedules and busyness, in evaluating perceived stress, wellbeing and other outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Residents in the following participating departments: departments of psychiatry, pediatrics, or neurology at MGH, medicine or psychiatry at NYU, or medicine or psychiatry at Cornell

Exclusion Criteria:

* Not a resident in the participating departments

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Change in burnout levels post intervention | change between baseline (July 2015), midpoint (week 25), to post intervention (week 52)
  Maslach Burnout Inventory (MBI), a validated 22-item self-report measure of professional burnout in human services. The MBI consists of 3 subscales of burnout: emotional exhaustion, depersonalization, and low sense of personal accomplishment.

SECONDARY OUTCOMES:
Change in perceived stress post intervention | change between baseline (July 2015), midpoint (week 25), to post intervention (week 52)
  Perceived Stress Scale (PSS-10)
Change in continuous physiologic data throughout intervention | change between baseline (July 2015), midpoint (week 25), to post intervention (week 52)
  Basis Peak Health Tracking device collects continuous physiologic data (heart rate, galvanized skin response, sleep duration and quality, exercise and actigraphy)
change in mindfulness post intervention | change between baseline (July 2015), midpoint (week 25), to post intervention (week 52)
  Cognitive and Affective Mindfulness Scale-Revised (CAMS-R)

CONTACTS AND LOCATIONS:
Overall Officials: John W Denninger, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Benson-Henry Institute for Mind Body Medicine, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Chaukos D, Zebrowski JP, Benson NM, Celik A, Chad-Friedman E, Teitelbaum A, Bernstein C, Cook R, Genfi A, Denninger JW. "One size does not fit all" - lessons learned from a multiple-methods study of a resident wellness curriculum across sites and specialties. BMC Med Educ. 2021 Nov 13;21(1):576. doi: 10.1186/s12909-021-02995-z. PMID 34774057